CLINICAL TRIAL: NCT00595348
Title: Korean Hereditary Breast Cancer Study
Acronym: KOHBRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Sung-Won Kim, Seoul National University Bundang Hospital, Surgery
Other Study IDs: KBCSG003; Sung-Won Kim, brca@korea.com
Record Dates: First submitted 2008-01-06; First posted 2008-01-16 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, Serum, plasma, Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. To evaluate the prevalence of BRCA1/2 mutation of breast cancer patients with family history of breast/ovarian cancer.
2. To evaluate the prevalence of BRCA1/2 mutation of breast cancer patients without family history, but high risk of hereditary cancer.
3. To evaluate the prevalence of BRCA1/2 mutation of family member of BRCA1/2 mutation.
4. To evaluate the prevalence of ovarian cancer of population of above 3 groups.

DETAILED DESCRIPTION:
1. To find founder mutation in Korean
2. To correlation prevalence with risk evaluation
3. To find risk factors concerning life style

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years old
* Agree to this study
* Breast cancer patient with family history of breast/ovarian cancer (1 subgroup)
* Breast cancer patient; young age (<40), bilateral, male, combined ovarian (2 subgroup)
* Family members with 1, 2 subgroups (3 subgroup)

Exclusion Criteria:

* Under 20 years old
* Unable to decide for oneself

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All Medical Center including personal breast clinic, general hospital, university hospital, cancer institute in Korea
Sampling Method: Non-Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2007-11; Primary Completion 2012-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Find out the prevalence of BRCA1/2 mutation of high risk breast cancer patients | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Won Kim, M.D, Ph.D., Principal Investigator — Department of Surgery, Breast & Endocrine Service, Seoul National University Bundang Hospital
Locations (1):
- Department of Surgery, Breast & Endocrine Service Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Ko KP, Kim SW, Ma SH, Park B, Ahn Y, Lee JW, Lee MH, Kang E, Kim LS, Jung Y, Cho YU, Lee B, Lin JH, Park SK. Dietary intake and breast cancer among carriers and noncarriers of BRCA mutations in the Korean Hereditary Breast Cancer Study. Am J Clin Nutr. 2013 Dec;98(6):1493-501. doi: 10.3945/ajcn.112.057760. Epub 2013 Oct 23. PMID 24153343
- [Derived] Han SA, Kim SW, Kang E, Park SK, Ahn SH, Lee MH, Nam SJ, Han W, Bae YT, Kim HA, Cho YU, Chang MC, Paik NS, Hwang KT, Kim SJ, Noh DY, Choi DH, Noh WC, Kim LS, Kim KS, Suh YJ, Lee JE, Jung Y, Moon BI, Yang JH, Son BH, Yom CK, Kim SY, Lee H, Jung SH; KOHBRA Research Group and the Korean Breast Cancer Society. The prevalence of BRCA mutations among familial breast cancer patients in Korea: results of the Korean Hereditary Breast Cancer study. Fam Cancer. 2013 Mar;12(1):75-81. doi: 10.1007/s10689-012-9578-7. PMID 23131904
- [Derived] Han SA, Park SK, Ahn SH, Lee MH, Noh DY, Kim LS, Noh WC, Jung Y, Kim KS, Kim SW; Korean Breast Cancer Study Group. The Korean Hereditary Breast Cancer (KOHBRA) study: protocols and interim report. Clin Oncol (R Coll Radiol). 2011 Sep;23(7):434-41. doi: 10.1016/j.clon.2010.11.007. Epub 2011 Apr 16. PMID 21497495